CLINICAL TRIAL: NCT01487863
Title: A Randomized, Open-label, Phase 2 Trial of Sipuleucel-T With Concurrent Versus Sequential Administration of Abiraterone Acetate Plus Prednisone in Men With Metastatic Castrate Resistant Prostate Cancer (mCRPC)
Brief Title: Concurrent vs. Sequential Sipuleucel-T & Abiraterone Treatment in Men With Metastatic Castrate Resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dendreon (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: P11-3
Record Dates: First submitted 2011-12-06; First posted 2011-12-08 (Estimated); Results first posted 2017-06-12 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Prostate Cancer Metastatic; Hormone Refractory Prostate Cancer; Castration-resistant Prostate Cancer
Keywords: prostate cancer; prostate; androgen independent prostate cancer (AIPC); androgen-independent; androgen independent; hormone insensitive; hormone-insensitive; prostate specific antigen (PSA); prostatic adenocarcinoma; hormone-refractory; hormone refractory; hormone refractory prostate cancer (HRPC); immune therapy; immunotherapy; vaccine; dendritic cells; antigen-presenting cells; antigen presenting cells; cancer vaccine; therapeutic vaccine; therapeutic cancer vaccine; recombinant; biological; biopharmaceutical; biotechnology; biotech; castration resistant prostate cancer (CRPC); castration-resistant prostate cancer (CRPC); castration-resistance; sipuleucel-T; abiraterone; prednisone; sequence; sequencing
MeSH Terms: conditions — Prostatic Neoplasms | interventions — sipuleucel-T; Abiraterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Concurrent Arm (Experimental): Subjects received sipuleucel-T concurrent with abiraterone acetate plus prednisone. Abiraterone acetate plus prednisone treatment started the next day after the first infusion of sipuleucel-T and continued for 26 weeks or until disease progression, unacceptable toxicity, or death, occurred.
  Interventions: Biological: sipuleucel-T; Drug: abiraterone acetate
- Sequential Arm (Experimental): Subjects received sipuleucel-T therapy followed by abiraterone acetate plus prednisone. Abiraterone acetate plus prednisone started at week 10 from the start of the first infusion of sipuleucel-T and continued for 26 weeks or until disease progression, unacceptable toxicity, or death, occurred.
  Interventions: Biological: sipuleucel-T; Drug: abiraterone acetate

INTERVENTIONS:
Biological: sipuleucel-T — Sipuleucel-T is an autologous cell product consisting of antigen presenting cells (APCs) loaded with PA2024, a recombinant fusion protein composed of prostatic acid phosphatase (PAP), linked to granulocyte-macrophage colony-stimulating factor (GM-CSF).
  Other Names: PROVENGE(R); APC8015
Drug: abiraterone acetate — Abiraterone acetate (1000 mg po QD) was administered in combination with prednisone (5 mg po BID) for a total of 26 weeks.
  Other Names: ZYTIGA(R)

SUMMARY:
The purpose of this study was to evaluate the impact of concurrent versus sequential administration of abiraterone acetate plus prednisone on the ability to manufacture sipuleucel-T (by assessing sipuleucel-T product parameters), and to assess the safety and efficacy of sipuleucel-T with concurrent or sequential administration of abiraterone acetate plus prednisone in men with metastatic castrate resistant prostate cancer.

DETAILED DESCRIPTION:
Subjects underwent screening procedures at the Screening Visit to ensure that they met the inclusion and exclusion criteria outlined in the protocol. Subjects were evaluated for eligibility criteria, and if eligible, were registered and randomized in a 1:1 into either the Concurrent Arm or the Sequential Arm.

Subjects in both arms underwent a standard 1.5 to 2.0 blood volume leukapheresis, followed approximately 3 days later by an intravenous (IV) infusion of sipuleucel-T. This process occurred at approximately 2-week intervals. A course of sipuleucel-T treatment comprised three infusions.

Following the first infusion, subjects were limited to a maximum of three total product failures for all subsequent infusions, due specifically to insufficient total nucleated cell (TNC) count and/or CD54 upregulation. These subjects received no further leukaphereses or sipuleucel-T infusions, but did receive abiraterone acetate plus prednisone per the schedule of the arm to which they were randomized. All subjects received a total of 26 weeks of abiraterone acetate plus prednisone therapy.

All immune monitoring (IM) endpoints were collected from all subjects who received at least one infusion. Cellular and serological immune responses were assessed for subjects in both arms. In both arms, IM blood samples were collected at baseline (screening); pre-leukapheresis 2 and 3; post-infusion 1, 2, and 3; and weeks 6, 10, 14, and 26, with the timing of IM visits based on the onset of treatment (Day 0). Day 0 was the day of the first infusion. Post-infusion blood draws occurred at 3 hours (allowable window 1-24 hours) after each infusion. If a subject received only one or two infusions, immune samples were still drawn at the scheduled time points based on the first infusion (Day 0). If the subject was not scheduled to undergo further leukapheresis, no other pre-leukapheresis procedures were conducted.

During the active follow-up phase, subjects were followed from registration through the Post-Treatment Visit (30-37 days post-last study treatment), or until disease progression, unacceptable toxicity, or death, whichever occurred first.

During the long-term follow-up (LTFU) phase, subjects were followed from the Post-Treatment Visit for up to 3 years from the date of registration/randomization. During the LTFU phase, only new treatment-related serious adverse event (SAE)s, cerebrovascular event (CVE)s (regardless of causality), the first anti-cancer therapy and first chemotherapy, and survival status were collected via a quarterly telephone call.

Overall survival was measured as the time from randomization until death over a 3-year period.

ELIGIBILITY:
Inclusion Criteria:

* histologically documented prostate cancer confirmed by a pathology report from prostate biopsy or radical prostatectomy specimen
* metastatic status as evidenced by imaging obtained </= 56 days prior to registration demonstrating bone metastasis or lymph node metastasis
* castrate resistant prostate cancer: castrate levels of testosterone (</= 50 ng/dL); evidence of disease progression concomitant with surgical or medical castration
* serum PSA >/= 2.0 ng/mL
* castrate levels of testosterone (</= 50 ng/dL) achieved via medical or surgical castration
* baseline Eastern Cooperative Oncology Group (ECOG) performance status of </= 1
* systolic blood pressure (BP) </= 140 mm Hg and diastolic BP </= 90 mm Hg at screening
* adequate baseline hematologic, renal, and liver functions
* must live in a permanent residence within a comfortable driving distance (round trip within one day) of the clinical trial site

Exclusion Criteria:

* the presence of known lung, liver, or brain metastases, malignant pleural effusions, or malignant ascites
* New York Heart Association Class III or IV heart failure
* any medical condition that may be compromised by increases in blood pressure, hypokalemia, or fluid retention
* Child-Pugh Class B or C hepatic insufficiency
* spinal cord compression, imminent long bone fracture, or any other condition likely to require radiation therapy and/or steroids for pain control
* known adrenalcortical insufficiency
* any medical contraindications to receiving prednisone
* prior treatment with sipuleucel-T
* previous treatment with abiraterone acetate (Zytiga(R)) or ipilimumab (Yervoy(TM))
* a requirement for systemic immunosuppressive therapy for any reason. Use of inhaled, intra-nasal, intra-articular, and topical steroids was allowed.
* treatment with any investigational vaccine or immunotherapy
* treatment with any chemotherapy prior to registration.
* a history of stage III or greater cancer, excluding prostate cancer. Basal or squamous cell skin cancers must have been adequately treated and the subject must be disease-free at the time of registration. Subjects with a history of stage I or II cancer must have been adequately treated and been disease-free for ≥ 3 years at the time of registration.
* myocardial infarction or ventricular or atrial arrhythmia within 6 months prior to registration
* ongoing anti-androgen withdrawal response.
* systemic steroid use within ≤ 60 days of registration
* treatment with denosumab (Xgeva(R) or Prolia (R)) within ≤ 3 months prior to registration
* positive test for human immunodeficiency virus (HIV) or human T cell lymphotrophic virus (HTLV) infections. Subjects with a positive test for hepatitis B or hepatitis C were allowed provided they meet the liver function test (LFT) criteria and have no signs of acute infection or active disease.
* treatment with any of the following medications or interventions within 28 days prior to registration: external beam radiation or major surgery requiring general anesthetic; saw palmetto; megestrol acetate (Megace(R)), diethylstilbestrol, and cyproterone; 5-alpha-reductase inhibitors (e.g. finasteride [Proscar(R)], dutasteride [Avodart(R)]); steroidal anti-androgen therapy; any other systemic therapy for prostate cancer, except for medical castration; treatment with any other investigational product for prostate cancer; substrates of CYP2D6 (e.g. including but not limited to thioridazine); inhibitors of CYP3A4 (e.g. including but not limited to ketoconazole, itraconazole, clarithromycin, nefazodone, telithromycin, and voriconazole); inducers of CYP3A4 (e.g. including but not limited to phenytoin, carbamazepine, rifampin, rifapentine, and phenobarbital)
* a requirement for treatment with opioid analgesics within 21 days prior to registration
* an active infection or infection requiring parenteral antibiotic therapy or causing fever within 7 days of registration
* any medical intervention, or other condition, or any other circumstance that, in the opinion of the Investigator or the Dendreon Medical Monitor, could compromise adherence with study requirements or otherwise compromise the study's objectives

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2011-12; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Israel, MD, Study Director — Valeant Pharmaceuticals North America LLC
Locations (21):
- United States (21):
  - UCSD Medical Center - La Jolla, La Jolla, California
  - Moores UCSD Cancer Center, La Jolla, California
  - Cancer Center Oncology Medical Group, La Mesa, California
  - UCSD Medical Center - Hillcrest, San Diego, California
  - Medical Oncology Associates - SD, San Diego, California
  - Sharp Rees-Stealy, San Diego, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - The Urology Center of Colorado, Denver, Colorado
  - Georgetown University Medical Center - Lombardi Cancer Center, Washington D.C., District of Columbia
  - Indiana University, Indianapolis, Indiana
  - Mid Atlantic Urology Associates, Mid Atlantic Clinical Research, Greenbelt, Maryland
  - GU Research Center, LLC, Omaha, Nebraska
  - NYU Clinical Cancer Center, NYU Langone Medical Center, New York, New York
  - The Mount Sinai Medical Center, New York, New York
  - Associated Medical Professionals of NY, PLLC, Oneida, New York
  - Associated Medical Professionals of New York, PLLC, Syracuse, New York
  - Providence Cancer Center Oncology and Hematology Care, Portland, Oregon
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology Associates, P.C., Nashville, Tennessee
  - Urology of Virginia, Virginia Beach, Virginia
  - Virginia Mason Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Antonarakis ES, Subudhi SK, Pieczonka CM, Karsh LI, Quinn DI, Hafron JM, Wilfehrt HM, Harmon M, Sheikh NA, Shore ND, Petrylak DP. Combination Treatment with Sipuleucel-T and Abiraterone Acetate or Enzalutamide for Metastatic Castration-Resistant Prostate Cancer: STAMP and STRIDE Trials. Clin Cancer Res. 2023 Jul 5;29(13):2426-2434. doi: 10.1158/1078-0432.CCR-22-3832. PMID 37058234

RESULTS

PARTICIPANT FLOW:
Groups:
- Concurrent Arm: Subjects received sipuleucel-T with concurrent abiraterone acetate plus prednisone. Abiraterone acetate plus prednisone treatment started the next day after the first infusion of sipuleucel-T and continued for 26 weeks or until disease progression, unacceptable toxicity, or death occurred.
  sipuleucel-T: Sipuleucel-T is an autologous cell product consisting of antigen presenting cells (APCs) loaded with PA2024, a recombinant fusion protein composed of prostatic acid phosphatase (PAP), linked to granulocyte-macrophage colony-stimulating factor (GM-CSF).
  abiraterone acetate: Abiraterone acetate (1000 mg po QD) was administered in combination with prednisone (5 mg po BID) for a total of 26 weeks.
- Sequential Arm: Subjects received sipuleucel-T therapy followed by abiraterone acetate plus prednisone. Abiraterone acetate plus prednisone started at week 10 from the start of the first infusion of sipuleucel-T and continued for 26 weeks or until disease progression, unacceptable toxicity, or death occurred.
  sipuleucel-T: Sipuleucel-T is an autologous cell product consisting of antigen presenting cells (APCs) loaded with PA2024, a recombinant fusion protein composed of prostatic acid phosphatase (PAP), linked to granulocyte-macrophage colony-stimulating factor (GM-CSF).
  abiraterone acetate: Abiraterone acetate (1000 mg po QD) was administered in combination with prednisone (5 mg po BID) for a total of 26 weeks.
Period: Overall Study
Arm/Group | Concurrent Arm | Sequential Arm
Started | 35 | 34
Subjects Randomized (Efficacy Analysis) | 35 | 34
Rcvd ≥1 Leukapheresis (Safety Analysis) | 35 | 34
Completed | 16 | 15
Not Completed | 19 | 19
Not completed — Death | 19 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Concurrent Arm | Sequential Arm | Total
Number analyzed (Participants) | 35 | 34 | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 11 | 24
  >=65 years | 22 | 23 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.7 (9.8) | 70.5 (10.15) | 70.1 (9.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 35 | 34 | 69
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 33 | 29 | 62
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 35 | 34 | 69
Weight [Mean (Standard Deviation); unit: Kg] | 94.22 (21.38) | 93.46 (16.29) | 93.85 (18.90)
Height [Mean (Standard Deviation); unit: Centimeters] | 176.10 (8.25) | 177.39 (8.06) | 176.73 (8.12)
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG Performance Status is a method used to assess the functional status of a patient. The scale ranges from 0-5. 0=Fully active, able to carry on all pre-disease performance without restriction; 1=Restricted in physically strenuous activity but ambulatory and able to carry out light or sedentary work; 2=Ambulatory, capable of all self-care but unable to carry out work activities. Up and about >50% of waking hour; 3=Capable of limited self-care, confined to bed or chair >50% of waking hours; 4=Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair; 5=Dead
  Participants
    ECOG 0=Fully Active; No restrictions | 28 | 26 | 54
    ECOG 1= Restricted Strenuous Activity | 7 | 8 | 15
Gleason Score [Count of Participants; unit: Participants] — Gleason score= prostate cancer grading system based on how tissue looks under a microscope. Scores range 2-10 and indicates how likely it is that a tumor will spread. A low score means the cancer tissue is similar to normal tissue and the tumor is less likely to spread. Gleason Score ≤ 6=the tumor is well differentiated, less aggressive and likely to grow more slowly;7=the tumor is moderately differentiated, moderately aggressive, and likely to grow but may not spread quickly;≥8=the tumor is poorly differentiated or undifferentiated, highly aggressive, and likely to grow faster and spread.
  Participants
    Gleason Score ≤ 6 | 5 | 5 | 10
    Gleason Score = 7 | 12 | 8 | 20
    Gleason Score ≥ 8 | 18 | 20 | 38
    Gleason Score - Missing Data | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Cumulative CD54 Upregulation Ratio Between the Cohorts.
Description: An analysis of variance model for the log transformed cumulative CD54 upregulation ratio (CD54 upregulation is the fold increase in the final product (FP) from buoyant density separations (BDS) step 65. BDS65 step refers to sample taken after both BDS77 and BDS65 but before ex vivo culture in the presence of antigen PA2024. FP refers to sample taken after ex vivo culture) that includes the antigen concentration cohort as the independent variable was performed. Subjects who received all 3 infusions were included.
Time Frame: Over the course of sipuleucel-T therapy (approximately 1 month)
Population: The efficacy population is defined as all randomized subjects. All the subjects in the efficacy population were analyzed according to the treatment that they were randomized to receive.
Measure: Mean (Standard Error); unit: Ratio ofCD54 molecules on BDS65:FP cells
Groups:
- Concurrent Arm: Subjects received sipuleucel-T concurrent with abiraterone acetate plus prednisone. Abiraterone acetate plus prednisone treatment started the next day after the first infusion of sipuleucel-T and continued for 26 weeks or until disease progression, unacceptable toxicity, or death occurred.
  sipuleucel-T: Sipuleucel-T is an autologous cell product consisting of antigen presenting cells (APCs) loaded with PA2024, a recombinant fusion protein composed of prostatic acid phosphatase (PAP), linked to granulocyte-macrophage colony-stimulating factor (GM-CSF).
  abiraterone acetate: Abiraterone acetate (1000 mg po QD) was administered in combination with prednisone (5 mg po BID) for a total of 26 weeks.
Arm/Group | Concurrent Arm | Sequential Arm
Number analyzed (Participants) | 35 | 34
Ratio ofCD54 molecules on BDS65:FP cells | 36.72 (2.32) | 41.61 (2.30)
Statistical Analysis 1: Comparison: Concurrent Arm vs Sequential Arm; Test type: Superiority; p = 0.2141, Wilcoxon (Mann-Whitney); Wilcoxon rank-sum test

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) and serious adverse events (SAEs) were recorded from registration until the Post-Treatment Visit (30-37 days after last study treatment). Only treatment-related AEs and cerebrovascular events (CVEs) ongoing at the Post-Treatment Visit, were followed until resolution, return to baseline or no further improvement was expected. After the Post-Treatment Visit, only new treatment-related SAEs and CVEs (regardless of causality) were collected and recorded as SAEs.
Arm/Group | Concurrent Arm | Sequential Arm
All-Cause Mortality (participants affected / at risk) | 19/35 | 19/34
Serious Adverse Events (participants affected / at risk) | 7/35 | 14/34
Other Adverse Events (participants affected / at risk) | 35/35 | 32/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Concurrent Arm (N=35) | Sequential Arm (N=34)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Disease Progression (General disorders) | 1 (1) | 2 (2)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 0 (0) | 1 (1)
Systemic Inflammatory Response Syndrome (General disorders) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Muscle Haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage Intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Obstructive Uropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureteric Obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertensive Crisis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Concurrent Arm (N=35) | Sequential Arm (N=34)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 7 (12)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (9) | 10 (12)
Paraesthesia Oral (Gastrointestinal disorders) | 8 (12) | 7 (14)
Constipation (Gastrointestinal disorders) | 4 (4) | 7 (8)
Diarrhoea (Gastrointestinal disorders) | 6 (7) | 3 (5)
Vomiting (Gastrointestinal disorders) | 3 (3) | 5 (6)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 3 (4)
Flatulence (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 10 (10) | 9 (17)
Oedema Periperal (General disorders) | 10 (12) | 5 (6)
Chills (General disorders) | 6 (9) | 8 (12)
Pyrexia (General disorders) | 7 (7) | 5 (8)
Pain (General disorders) | 1 (1) | 7 (8)
Influenza Like Illness (General disorders) | 1 (1) | 5 (8)
Asthenia (General disorders) | 3 (3) | 2 (2)
Gait Disturbance (General disorders) | 1 (1) | 3 (3)
Chest Pain (General disorders) | 0 (0) | 3 (4)
Oedema (General disorders) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (3)
Urinary Tract Infection (Infections and infestations) | 3 (3) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2)
Influenza (Infections and infestations) | 0 (0) | 2 (2)
Oral Herpes (Infections and infestations) | 0 (0) | 2 (2)
Citrate Toxicity (Injury, poisoning and procedural complications) | 3 (8) | 6 (12)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 2 (3)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Blood Alkaline Phosphatase Increased (Investigations) | 0 (0) | 3 (3)
Blood Urea Increased (Investigations) | 0 (0) | 2 (2)
Heart Rate Irregular (Investigations) | 2 (2) | 0 (0)
Weight Decreased (Investigations) | 0 (0) | 2 (2)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 17 (22) | 9 (14)
Back Pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 10 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 7 (9)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 8 (11)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 3 (3)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 4 (6) | 2 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (5) | 3 (5)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Paraesthesia (Nervous system disorders) | 5 (6) | 6 (8)
Headache (Nervous system disorders) | 5 (5) | 5 (6)
Dizziness (Nervous system disorders) | 2 (2) | 6 (9)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 4 (4)
Tremor (Nervous system disorders) | 1 (1) | 3 (3)
Dysgeusia (Nervous system disorders) | 1 (1) | 2 (3)
Syncope (Nervous system disorders) | 0 (0) | 2 (3)
Anxiety (Psychiatric disorders) | 3 (3) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 3 (3)
Depression (Psychiatric disorders) | 0 (0) | 3 (4)
Pollakiuria (Renal and urinary disorders) | 2 (2) | 3 (3)
Haematuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Dysuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 2 (3)
Gynaecomastia (Reproductive system and breast disorders) | 2 (2) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 7 (10)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (7)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 4 (6) | 4 (5)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Hot Flush (Vascular disorders) | 5 (5) | 3 (3)
Hypertension (Vascular disorders) | 4 (4) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the Study will be published and/or presented in an integrated manner reflecting the results observed across all participating centers. Accordingly, decisions on timing and content of publications and presentations relating to the Study will be coordinated by Dendreon in communication with institutions contributing patients to the Study.